CLINICAL TRIAL: NCT04292444
Title: Disentangling Effects of Oxytocin on Cognitive and Reactive Fear and the Moderating Role of the Receptor for Advanced Glycation End-products
Brief Title: Effects of Oxytocin on Cognitive and Reactive Fear
Acronym: RAGE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, Professor for Psychiatry, University of Oldenburg
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RAGE
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Oxytocin
Keywords: fMRI; receptor for advanced glycation end-products (RAGE); fear; 7T MRI

STUDY DESIGN:
Intervention Model Description: The study is designed as a double-blind, within-subject, placebo-controlled, non-clinical trial and will involve healthy male participants (n = 60), who will be scanned twice in a randomized order after a single dose of intranasal OXT (24 IU) or placebo. Furthermore participants will be pre-stratified based on a RAGE polymorphism (-374 T/A: rs1800624; n = 30 with TT alleles and n = 30 with TA/AA alleles).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAGE polymorphism (TT) (Experimental): 30 participants with the RAGE polymorphism (-374 T/A: rs1800624; TT) will be selected and scanned twice.
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo
- RAGE polymorphism (TA/AA) (Experimental): 30 participants with the RAGE polymorphism (-374 T/A: rs1800624; TA/AA) will be selected and scanned twice.
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — Intranasal administration of 24 International Units oxytocin 30 minutes before the start of the tasks.
Drug: Placebo — The placebo nasal sprays contain identical ingredients except for the peptide itself (30 minutes before the start of the tasks).

SUMMARY:
The study examines the (sub)regional specificity of anxiolytic oxytocin (OXT) effects on emotional face processing and reactive and cognitive fear. Preliminary data indicate that the Receptor for Advanced Glycation End Products (RAGE) may regulate oxytocin transport into the brain. Thus, the study aims to replicate previous observations of oxytocin effects on the processing of fearful faces in the centro-medial amygdala and to assess whether a RAGE polymorphism (-374 T/A: rs1800624; TT vs. TA/AA), that has been shown to alter transcriptional activity, modulates anxiolytic OXT effects.

DETAILED DESCRIPTION:
So far, no study examined selective oxytocin (OXT) effects on reactive (midbrain periaqueductal gray (PAG), central amygdala (CeA), hypothalamus, and the midcingulate cortex (MCC)) and cognitive fear (ventromedial prefrontal cortex (vmPFC), posterior cingulate cortex (PCC), hippocampus, and basolateral amygdala) and the reward system (striatum) with high spatial resolution. Previous studies showed that 7T functional magnetic resonance imaging (fMRI) results in a higher spatial resolution and specificity than 3T MRI in these brain regions and would thus allow for a more detailed characterization of the neural effects.

To disentangle (sub)region-specific effects of OXT on task-related activations of the cingulate structures, the amygdala, the striatum, PAG and VMPFC, the investigators plan to acquire ultra-high field 7T fMRI data from healthy male participants while they perform (i) an emotional face matching task and (ii) a flight initiation distance (FID) task involving fast- or slow-attacking virtual predators that elicit distinct activations in the reactive and cognitive fear circuits. Furthermore, participants will be pre-stratified depending on RAGE polymorphisms to elucidate possible RAGE-related differential OXT effects.

ELIGIBILITY:
Inclusion Criteria:

* RAGE polymorphism (-374 T/A: rs1800624; TT vs. TA/AA)
* healthy male volunteers
* right handed

Exclusion Criteria:

* current psychiatric illness
* current psychiatric medication or psychotherapy
* MRI contraindication (e.g. metal in body, claustrophobia)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Neural substrates of emotion processing, measured via blood-oxygen-level dependent (BOLD) signal in the amygdala and striatum | 30 minutes after nasal spray administration
  Functional magnetic resonance imaging will be performed to measure the BOLD signal in response to emotional face stimuli. The investigators specifically plan to investigate neural responses to emotional faces in amygdala and striatal subregions. The BOLD signal in response to fearful faces relative to neutral faces and happy faces relative to neutral will be compared between the oxytocin and placebo sessions. To examine effects of the Receptor for Advanced Glycation End Products (RAGE), analyses of variance (ANOVAs) with the between subjects factor RAGE polymorphism (-374 T/A: rs1800624; TT vs. TA/AA) will be conducted on the second level. For analyses of fMRI data, default procedures of the software SPM12 will be adapted for ultra-high-field imaging. The family-wise error rate will be used to correct p-values for multiple comparisons and p < .05 will be considered significant.
Neural responses in the flight initiation distance (FID) task | 45 minutes after nasal spray administration
  Functional magnetic resonance imaging will be performed to measure the blood-oxygen-level dependent (BOLD) signal in a flight initiation distance (FID) task, involving fast-, medium- and slow-attacking virtual predators that elicit distinct activations in the reactive and cognitive fear circuits. BOLD signals to different predator velocities will be analyzed. Analyses will focus on regions-of-interest associated with the processing of cognitive fear (vmPFC, PCC, hippocampus, and basolateral amygdala) and reactive fear (midbrain PAG, central amygdala, hypothalamus, and the MCC) and the reward system (striatum). To examine effects of the Receptor for Advanced Glycation End Products (RAGE), ANOVAs with the between-subject factor RAGE polymorphism (-374 T/A: rs1800624; TT vs. TA/AA) will be conducted on the 2nd level. For the fMRI data, default procedures of the software SPM12 will be adapted for ultra-high-field imaging.
Flight distance and difficulty ratings in the flight initiation distance (FID) task | 45 minutes after nasal spray administration
  Behavioral data of the FID task (flight distance and difficulty ratings ) will be analyzed using mixed ANOVAs in the software SPSS with treatment (oxytocin vs. placebo) as within-subject factor and RAGE polymorphism (TT vs. TA/AA) as between-subject factor. Post-hoc t-tests will be Bonferroni-corrected. Behavioral data will be correlated with fMRI data of the FID task.

SECONDARY OUTCOMES:
Oxytocin concentration in blood plasma | 10 minutes before nasal spray administration and 75 minutes after nasal spray administration
  Blood samples will be collected before and after the nasal spray administration to assess changes in oxytocin concentrations. Oxytocin concentrations will be analyzed using mixed ANOVAs in SPSS with time (pre vs. post) and treatment (oxytocin vs. placebo) as within-subject factors and RAGE polymorphism (TT vs. TA/AA) as between-subject factor.
Concentration of receptor for advanced glycation endproducts (extracellular domain) in blood plasma | 10 minutes before nasal spray administration
  Blood samples will be collected before the nasal spray administration to assess the RAGE (extracellular domain) concentration in blood plasma.
  RAGE concentrations will be compared between RAGE polymorphisms (TT vs. TA/AA) with independent t-tests. Furthermore, the investigators plan to examine if the RAGE concentration moderates the effects of oxytocin on primary and secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Hurlemann, MSc, MD, PhD, Principal Investigator — University of Oldenburg
Locations (1):
- Department of Psychiatry and Medical Psychology, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hahn A, Kranz GS, Seidel EM, Sladky R, Kraus C, Kublbock M, Pfabigan DM, Hummer A, Grahl A, Ganger S, Windischberger C, Lamm C, Lanzenberger R. Comparing neural response to painful electrical stimulation with functional MRI at 3 and 7 T. Neuroimage. 2013 Nov 15;82:336-43. doi: 10.1016/j.neuroimage.2013.06.010. Epub 2013 Jun 12. PMID 23769917
- [Background] Hudson BI, Stickland MH, Futers TS, Grant PJ. Effects of novel polymorphisms in the RAGE gene on transcriptional regulation and their association with diabetic retinopathy. Diabetes. 2001 Jun;50(6):1505-11. doi: 10.2337/diabetes.50.6.1505. PMID 11375354
- [Background] Qi S, Hassabis D, Sun J, Guo F, Daw N, Mobbs D. How cognitive and reactive fear circuits optimize escape decisions in humans. Proc Natl Acad Sci U S A. 2018 Mar 20;115(12):3186-3191. doi: 10.1073/pnas.1712314115. Epub 2018 Mar 5. PMID 29507207
- [Background] Yamamoto Y, Liang M, Munesue S, Deguchi K, Harashima A, Furuhara K, Yuhi T, Zhong J, Akther S, Goto H, Eguchi Y, Kitao Y, Hori O, Shiraishi Y, Ozaki N, Shimizu Y, Kamide T, Yoshikawa A, Hayashi Y, Nakada M, Lopatina O, Gerasimenko M, Komleva Y, Malinovskaya N, Salmina AB, Asano M, Nishimori K, Shoelson SE, Yamamoto H, Higashida H. Vascular RAGE transports oxytocin into the brain to elicit its maternal bonding behaviour in mice. Commun Biol. 2019 Feb 25;2:76. doi: 10.1038/s42003-019-0325-6. eCollection 2019. PMID 30820471
- [Background] Hariri AR, Tessitore A, Mattay VS, Fera F, Weinberger DR. The amygdala response to emotional stimuli: a comparison of faces and scenes. Neuroimage. 2002 Sep;17(1):317-23. doi: 10.1006/nimg.2002.1179. PMID 12482086
- See also: Neuromodulation of Emotion (NEMO) Research Group — http://renehurlemann.squarespace.com/welcome/